CLINICAL TRIAL: NCT02999308
Title: Hematology Oncology Center
Brief Title: A Clinical Phenotype Based Individualized Prophylaxis in Chinese Hemophilia A Children
Acronym: CHIPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Runhui WU, Chief doctor, Beijing Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIPS
Record Dates: First submitted 2016-09-01; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Haemophilia
Keywords: haemophilia; prophylaxis; children
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental)
  Interventions: Other: Observe the patient's condition and then change the regimen

INTERVENTIONS:
Other: Observe the patient's condition and then change the regimen — The patients will be assessed every 3 months and the treatment regimen will be modified by the result of assessment.

SUMMARY:
In the past, due to economic and medical resource constraints, the hemophilia comprehensive care in China was suboptimal. The BCH data of both retrospective and prospective studies reveals that for 4-6y and 6-9y patients with severe hemophilia respectively: 45% and 82% of the patients have suffered from joint bleeding, with mean AJBR of 4.18 and 4.95; and 24.2% and 33.3% of them with AJBR>10 times, led to arthropathies and made their quality of life be heavy affected. Now, with the development of economy and medical science in China, prophylaxis regimens have been initiated in more and more children with hemophilia. Considering the difference between prophylaxis regimens, the frequency of joint bleeding was reduced significantly, the quality of life of hemophilia kids improved. An assessment scoring system for the appropriate validation of individualized prophylaxis treatment regimens are urgently needed.

Before, the most important assessed indication for hemophilia prophylaxis was the frequency of joint bleeding. But increasing evidences are showing that there is a discrepancy between real joint damage and joint bleeding frequency. The single indicator of joint bleeding frequency is not sufficient to evaluate the joint status of hemophilia children.

Under the World Health Organization's ICF guidelines, the assessment scoring system for selecting prophylaxis for children with hemophilia should include the tools currently available for assessment of structure/function of the joint, patient activities and patient participation in hemophilia healthcare. According to ICF of WHO, the most common bleeding parts are elbows, knees and ankles, therefore the assessment of children with hemophilia should include the evaluation of the structure, the function of these 6 Index joints, the capacity of activities and the capacity of participation of children. These will constitute a comprehensive hemophilia evaluation system.

In China, exploration of the optimal and individualized prophylaxis regimen is urgent, and the comprehensive evaluation system should include joint structure and function, body's activities and individual participation, thus may be more appropriate for the individualized prophylaxis for Chinese children with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

1. Severe hemophilia A (FVIII: C<2%),
2. Age 1-7y
3. Historical bleeding in any knee, elbow and ankle joint (s),
4. >50 EDs irrespective of FVIII product, including human coagulate factor and recombinant factor VIII
5. No inhibitor present or history/family history,
6. On-demand or low-dose prophylaxis (the dose per kg.week less or as Step 1 prophylaxis regimens factor consumption)
7. Regular clinical visit with accessible data,
8. Informed consent will be obtained from patient legal guardians before the enrollment.

Exclusion Criteria:

* 1. Other bleeding disorders or systemic disorders, or don't fit for enrollment according to the investigator, 2. FVIII inhibitor development:>0.6 BU (confirmed by two separate tests), 3. Unable to follow the protocol or refuse to continue the participation.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of Ultrasound HEAD-US score of index joints | baseline,3 months, 6 months,9 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wu Runhui, MD, PhD, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Berntorp E, Boulyjenkov V, Brettler D, Chandy M, Jones P, Lee C, Lusher J, Mannucci P, Peak I, Rickard K, et al. Modern treatment of haemophilia. Bull World Health Organ. 1995;73(5):691-701. PMID 8846496
- [Result] Nilsson IM, Berntorp E, Lofqvist T, Pettersson H. Twenty-five years' experience of prophylactic treatment in severe haemophilia A and B. J Intern Med. 1992 Jul;232(1):25-32. doi: 10.1111/j.1365-2796.1992.tb00546.x. PMID 1640190